CLINICAL TRIAL: NCT05621629
Title: Strategies for Predicting the Efficacy of Sacral Nerve Stimulation With Pelvic Floor Rehabilitation in the Management of Fecal Incontinence After Surgery of Anorectal Malformation.
Brief Title: Management of FI After Surgery of ARM
Status: Completed | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Shucheng Zhang, Professor, Shengjing Hospital
Other Study IDs: A333-3
Record Dates: First submitted 2022-08-28; First posted 2022-11-18 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Fecal Incontinence; Childhood ALL; Anorectal Malformations
MeSH Terms: conditions — Fecal Incontinence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anorectal Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The posterior sagittal approach to anorectal malformation (ARM) has radically changed the outcome of these patients, improving the preservation of anal sphincters, owing to their anatomical identification. However, in long term follow-up, fecal incontinence and severe constipation remain the most frequent and disabling postoperative clinical problems, having a significant influence on quality of life. Current therapeutic measures for Fecal Incontinence include biofeedback, sacral nerve stimulation, radiofrequency energy delivery, surgical treatment and sphincter replacement. Biofeedback combined with SNS has achieved satisfactory results. However, not all patients have an improvement in their weakened anal sphincter and achieve acceptable continence.

A detailed assessment of anorectal sphincter morphology and function can predict therapeutic outcome. Magnetic resonance imaging(MRI) can help to judge the anal atresia type, to display the presence and running of the fistula, and to show the nature of anal sphincter, such as the shape, thickness, directions and position of the anal sphincter complex and location in the pelvic floor and other systems malformations, finally to provide a reliable diagnostic basis for surgical program and prognostic assessment. High-resolution anorectal manometry (HR-ARM) is the latest internationally recognized examination for the evaluation of anorectal function. A standardised protocol of HR-ARM can characterise FI from dyssynergic or other neuromuscular and sensory problems. As a result, HR-ARM provides a more appropriate management in patients with FI. In order to assess whether patients with fecal incontinence should choose biofeedback therapy, our study included children with FI after anorectal malformation, and combined HR-ARM and MR to predict the efficacy of sacral nerve stimulation and pelvic floor rehabilitation.

DETAILED DESCRIPTION:
The posterior sagittal approach to anorectal malformation (ARM) has radically changed the outcome of these patients, improving the preservation of anal sphincters, owing to their anatomical identification. However, in long term follow-up, fecal incontinence and severe constipation remain the most frequent and disabling postoperative clinical problems, with an important impact on quality of life. A cluster of physical and psychological problems appear in pediatric patients, including repeated infections, skin ulcer and scar, social anxiety disorder, behavioral problems, self-abasement or isolation and other problems, which cause children full of guilt and embarrassment and increase the risk of bullying.

Current therapeutic measures for FI include biofeedback, sacral nerve stimulation, radiofrequency energy delivery , surgical treatment, and sphincter replacement. Zhengwei Yuan et al. conducted a follow-up study on 31 patients with FI after ARM, and confirmed that biofeedback combined with SNS has a good effect on patients with FI after ARM. However,not all patients improve their impaired anal sphincter and acquire satisfactory continence. A lot of time and treatment costs are wasted. Therefore, it is necessary to clarify the indications for the application of biofeedback combined with SNS.

Severity of ARM affects the degree of development of internal and external anal sphincters. A detailed assessment of anorectal sphincter morphology and function can predict therapeutic outcome. In clinical practice, endoanal ultrasound and endoanal magnetic resonance imaging (MRI) are the main imaging modalities for the anatomical assessment of the anal sphincter complex. Sphincter MR is more suitable for observing the nature of the anal sphincter such as the shape, thickness, directions, and position of the anal sphincter complex and its location on the pelvic floor. MR examination has a high clinical value in the diagnosis of ARM. It can help determine the anal atresia type, display the presence and running of the fistula, evaluate the perianal muscle development and other systems' malformations, and finally provide a reliable diagnostic basis for surgical program and prognostic assessment. The role of MR is similar to that of EUS in some aspects. However, the sphincter MRI can clearly demonstrate the sphincter pattern, the position of the sphincter on the pelvic floor, and several indicators that cannot be detected by EUS. High-resolution anorectal manometry (HR-ARM) is the latest internationally recognized examination for the evaluation of anorectal function. A standardised protocol of HR-ARM can characterise FI from dyssynergic or other neuromuscular and sensory problems.Therefore, HR-ARM provides a more appropriate management in patients with FI. The anorectal manometry is a functional study that can evaluate the potential for muscular sphincterial recovery after BFB; the assessment derives greater benefit also from a morphological evaluation (MRI) in particular when the manometry is unfavorable.

The study included children with FI after ARM, and the investigators combined HR-ARM and MR to predict the efficacy of sacral nerve stimulation and pelvic floor rehabilitation to determine whether patients with fecal incontinence should choose biofeedback therapy.

ELIGIBILITY:
Inclusion Criteria:

1.4-18 years old; 2.The voluntary or involuntary defecation in an inappropriate place during children's developmental age of 4 years or above; 3.Anorectal malformation, anal reconstruction surgery was performed immediately after birth, and at least two courses of biofeedback combined with SNS were experienced 4.Clinical data are complete and sphincter MR and anorectal manometry have been done.

Exclusion Criteria:

1. Congenital and/or acquired intestinal diseases, such as congenital or severe secondary megacolon, intestinal stenosis, polyps, Crohn's disease, tuberculosis, inflammation, and tumours;
2. Neurological diseases, such as brain and spinal cord diseases, genetic metabolic diseases;
3. Psychosocial and behavioural diseases, and other systemic diseases;
4. Refused to MR and biofeedback combined with SNS.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Fecal Incontinence after surgery of Anorectal Malformation
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Average anal resting pressure | Baseline (Before treatment)
  Average maximum pressure (mm Hg) over the functional anal canal length during the 30-s period of rest
Maximum anal squeeze pressure | Baseline (Before treatment)
  Maximum pressure (mm Hg) sustained over the duration of the 5-s squeeze maneuver
Functional anal canal length (FACL) | Baseline (Before treatment)
  Length of anal canal (cm) in which pressure exceeded rectal pressure by >5 mm Hg
Thickness of the external anal sphincter | Baseline (Before treatment)
  Three measurements were made laterally for the external anal sphincter where the muscle appeared thickest during sphincter MRI , and an average value was determined.
Thickness of the internal anal sphincter | Baseline (Before treatment)
  The thickness of the internal anal sphincter was measured three times at a centimeter above the external sphincter during sphincter MRI.
Whether the rectum passes through the center of puborectalis | Baseline (Before treatment)
  Whether the rectum crosses the center of the puborectalis muscle on sphincter MRI.
Pena's questionnaires score after treatment | at the end of 4-weeks Biofeedback combined with SNS treatment
  select the pena questionnaire to assess bowel function in patients with fecal incontinence after anorectal malformation after treatment.
Pena's questionnaires score before treatment | Baseline (Before treatment)
  select the pena questionnaire to assess bowel function in patients with fecal incontinence after anorectal malformation before treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

REFERENCES:
- [Background] Loganathan AK, Mathew AS, Kurian JJ. Assessment of Quality of Life and Functional Outcomes of Operated Cases of Hirschsprung Disease in a Developing Country. Pediatr Gastroenterol Hepatol Nutr. 2021 Mar;24(2):145-153. doi: 10.5223/pghn.2021.24.2.145. Epub 2021 Mar 4. PMID 33833970
- [Background] Rajindrajith S, Devanarayana NM, Thapar N, Benninga MA. Functional Fecal Incontinence in Children: Epidemiology, Pathophysiology, Evaluation, and Management. J Pediatr Gastroenterol Nutr. 2021 Jun 1;72(6):794-801. doi: 10.1097/MPG.0000000000003056. PMID 33534361
- [Background] Bharucha AE, Rao SSC, Shin AS. Surgical Interventions and the Use of Device-Aided Therapy for the Treatment of Fecal Incontinence and Defecatory Disorders. Clin Gastroenterol Hepatol. 2017 Dec;15(12):1844-1854. doi: 10.1016/j.cgh.2017.08.023. Epub 2017 Aug 22. PMID 28838787
- [Background] Divarci E, Ergun O. General complications after surgery for anorectal malformations. Pediatr Surg Int. 2020 Apr;36(4):431-445. doi: 10.1007/s00383-020-04629-9. Epub 2020 Feb 21. PMID 32086570
- [Background] Sulkowski JP, Nacion KM, Deans KJ, Minneci PC, Levitt MA, Mousa HM, Alpert SA, Teich S. Sacral nerve stimulation: a promising therapy for fecal and urinary incontinence and constipation in children. J Pediatr Surg. 2015 Oct;50(10):1644-7. doi: 10.1016/j.jpedsurg.2015.03.043. Epub 2015 Mar 26. PMID 25858097
- [Background] Brown HW, Dyer KY, Rogers RG. Management of Fecal Incontinence. Obstet Gynecol. 2020 Oct;136(4):811-822. doi: 10.1097/AOG.0000000000004054. PMID 32925633
- [Background] Bjorsum-Meyer T, Christensen P, Baatrup G, Jakobsen MS, Asmussen J, Qvist N. Magnetic resonance imaging of the anal sphincter and spine in patients with anorectal malformations after posterior sagittal anorectoplasty: a late follow-up cross-sectional study. Pediatr Surg Int. 2021 Jan;37(1):85-91. doi: 10.1007/s00383-020-04774-1. Epub 2020 Nov 3. PMID 33141917
- [Background] Bischoff A, de La Torre L, Pena A. Comparative effectiveness of imaging modalities for preoperative assessment of anorectal malformation in the pediatric population. J Pediatr Surg. 2020 Feb;55(2):354. doi: 10.1016/j.jpedsurg.2019.09.078. Epub 2019 Oct 27. No abstract available. PMID 31718867
- [Background] Ambartsumyan L, Shaffer M, Carlin K, Nurko S. Comparison of longitudinal and radial characteristics of intra-anal pressures using 3D high-definition anorectal manometry between children with anoretal malformations and functional constipation. Neurogastroenterol Motil. 2021 Feb;33(2):e13971. doi: 10.1111/nmo.13971. Epub 2020 Sep 9. PMID 32902923
- [Background] Bjorsum-Meyer T, Christensen P, Jakobsen MS, Baatrup G, Qvist N. Correlation of anorectal manometry measures to severity of fecal incontinence in patients with anorectal malformations - a cross-sectional study. Sci Rep. 2020 Apr 7;10(1):6016. doi: 10.1038/s41598-020-62908-w. PMID 32265467
- [Background] Yates G, Friedmacher F, Cleeve S, Athanasakos E. Anorectal manometry in pediatric settings: A systematic review of 227 studies. Neurogastroenterol Motil. 2021 Apr;33(4):e14006. doi: 10.1111/nmo.14006. Epub 2020 Oct 28. PMID 33118295
- [Background] Koppen IJN, Vriesman MH, Saps M, Rajindrajith S, Shi X, van Etten-Jamaludin FS, Di Lorenzo C, Benninga MA, Tabbers MM. Prevalence of Functional Defecation Disorders in Children: A Systematic Review and Meta-Analysis. J Pediatr. 2018 Jul;198:121-130.e6. doi: 10.1016/j.jpeds.2018.02.029. Epub 2018 Apr 12. PMID 29656863
- [Background] Brisighelli G, Macchini F, Consonni D, Di Cesare A, Morandi A, Leva E. Continence after posterior sagittal anorectoplasty for anorectal malformations: comparison of different scores. J Pediatr Surg. 2018 Sep;53(9):1727-1733. doi: 10.1016/j.jpedsurg.2017.12.020. Epub 2017 Dec 27. PMID 29370894
- [Derived] Shen ZY, Zhang Y, Tao CH, Wang DJ, Zhang ZB, Zhang SC. A Predictive Model to Identify the Effects of Transcutaneous Sacral Nerve Stimulation With Pelvic Floor Exercises in Fecal Incontinence After Surgery for Anorectal Malformation. Am J Gastroenterol. 2024 Jan 1;119(1):191-199. doi: 10.14309/ajg.0000000000002544. Epub 2023 Oct 3. PMID 37787428